CLINICAL TRIAL: NCT05748145
Title: Preoperative Treatment With Metronidazole to Evaluate the Efficacy in Reducing Fusobacterium Nucleatum Tumor Colonization in Patients With Colorectal Cancer (CRC): a Proof-of-concept Trial
Brief Title: Metronidazole as Preoperative Therapy in CRC / FusoMetro-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oncology Institute of Southern Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FusoMetro-001
Record Dates: First submitted 2023-01-26; First posted 2023-02-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Proof of concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metronidazole treated arm (Experimental): Administration of Metronidazole for 10 days prior to surgery in CRC patients
  Interventions: Drug: Metronidazole Oral

INTERVENTIONS:
Drug: Metronidazole Oral — Metronidazole will be administered per os at 500 mg x 3/day, for 10 days prior to surgery.

SUMMARY:
The proposed proof-of concept trial aims at determining the effectiveness of metronidazole in decreasing the Fusobacterium nucleatum load in tissues and possibly on its detrimental effects on tumor cells and tumor microenvironment.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is among the most frequent tumor types and is a leading cause of cancer-related death worldwide. Surgery represents the first therapeutic option, whereas advanced cases are usually treated by established chemotherapy protocols, yet with variable response rates.

Mechanisms underlying unresponsiveness are still largely unclear. Recently, the gut microbiota, consisting of trillions of microorganisms, which populate the gastrointestinal tract, has also been implicated in chemo-resistance.

Defined bacterial species have been reported to be associated with CRC. In particular, Fusobacterium nucleatum (F.n.), a commensal bacterium of the oral cavity, is enriched in CRC tissues and its abundance appears to be associated with reduced patient survival.

In experimental models F.n. promotes CRC cell proliferation and reduces tumor responsiveness to 5-fluorouracil (5-FU). Furthermore, it suppresses tumor infiltration by immune cells associated with improved prognosis.

Administration of metronidazole effectively reduces F.n. load and overall tumor growth in animal models.

However, its efficacy in reducing F.n. loads in human CRC has not been verified so far.

The proposed proof-of concept trial aims at determining the effectiveness of metronidazole in decreasing the F.n. load in tissues and possibly on its detrimental effects on tumor cells and tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration.
* Age ≥ 18 years old
* Untreated, primary colorectal adenocarcinoma (> 15 cm from the anal verge)
* Colonoscopy with endoscopic biopsy for disease confirmation and correlative studies.
* Candidates for surgical resection prior to administration of any therapy.

Exclusion Criteria:

* Insufficient material on the tissue biopsy to be left in the archives of the Cantonal Institute of Pathology for further evaluations/analyses
* Known prior history of hypersensitivity to metronidazole or other nitroimidazole derivatives
* Oral or parenteral antibiotic therapy within the six weeks prior to enrolment
* Emergency surgery (planned within less than 14 days), where no opportunity to administer preoperative oral antibiotics exists
* Other malignant disease within 5 years prior to study enrollment, except basocellular or squamous skin cancer and carcinoma in situ cervices uteri
* Any previous anticancer treatment prior resection
* Women who are pregnant or breast feeding
* Fertile women or men who do not use safe contraception during the study period
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Inability to consent and follow the procedures of the study e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment, affect patient compliance or place the patient at high risk from treatment-related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of metronidazole on F.n. loads in CRC tissues. | 12 (+ 3) days after surgery
  F.n. load assessed by qRT-PCR analysis in excised tumor tissues upon antibiotic treatment, as compared to corresponding diagnostic biopsies prior to treatment.

SECONDARY OUTCOMES:
Potential effects of metronidazole on the expression of immune cell markers in CRC tissue samples | 12 (+ 3) days after surgery
  Expression of multiple immune cell markers will be assessed in tissue samples by immunohistochemistry and immunofluorescence. Number of positive cells/mm2 will be evaluated.
Potential effects of metronidazole on the expression of autophagy markers in CRC tissue samples | 12 (+ 3) days after surgery
  Expression of multiple autophagy signaling elements will be assessed in tissue samples by immunohistochemistry and immunofluorescence. Number of positive cells/mm2 will be evaluated.
Potential effects of metronidazole on microbiome | 12 (+ 3) days after surgery
  Differences in community diversity and/or abundance of specific bacterial taxa between the tumor-associated microbiome prior to or after antibiotic treatment.
Potential effects of metronidazole on the intestinal metabolic profile | 12 (+ 3) days after surgery
  Measurement of changes in the biosynthesis pathways of intestinal bacteria by comparing the gut metabolic profile before and after antibiotic treatment. Fold changes in the abundance of bacterial metabolites will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Southern Switzerland, Bellinzona, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided